CLINICAL TRIAL: NCT03090919
Title: The INFUSE Trial - Intervening With Platelet Transfusions in Sepsis
Acronym: INFUSE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Susan Smyth (Other)
Responsible Party: Sponsor-Investigator, Susan Smyth, Principle Investigators, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0784-F6A
Record Dates: First submitted 2017-01-24; First posted 2017-03-27 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Sepsis; Thrombocytopenia
MeSH Terms: conditions — Sepsis; Thrombocytopenia | interventions — Platelet Transfusion; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to recieve either a platelet transfusion or a saline transfusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator): Subjects randomized to the Saline arm will receive 250cc of physiological saline.
  Interventions: Other: Saline
- Platelet transfusion (Experimental): Subjects randomized to platelet transfusion will receive a unit of platelets (~250cc in volume).
  Interventions: Biological: Platelet transfusion

INTERVENTIONS:
Biological: Platelet transfusion
  Arms: Platelet transfusion
Other: Saline
  Arms: Saline

SUMMARY:
Sepsis is life-threatening and dysregulated response to infection that results in endothelial activation and dysfunction that leads to systemic microvascular leak and multiple-organ failure. This study will identify patients that have sepsis with thrombocytopenia and randomize them to receive a unit of platelets or an equivalent volume of saline.

DETAILED DESCRIPTION:
Sepsis is life-threatening and dysregulated response to infection that results in endothelial activation and dysfunction that leads to systemic microvascular leak and multiple-organ failure. Emerging evidence indicates that platelets occupy a central role in maintaining the balance between vascular health and the response to environmental changes and vascular injury. Platelets are essential for vascular development and required for normal endothelial integrity. Platelets also function at the interface between thrombosis and inflammation. This study will identify patients that have sepsis with thrombocytopenia and randomize them to receive a unit of platelets or an equivalent volume of saline.

Our overall hypotheis is that normal platelet function is required to maintain vascular integrity and can be at least partially restored over the first 24 hours by platelet transfusion in septic patients with thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria

* Provision of informed consent prior to any study specific procedures
* Female and/or male, age >18 years
* Diagnosis of sepsis based on the Third International Consensus Definitions for Sepsis and Septic Shock
* Platelet count ≤ 50,000/μL

Exclusion Criteria

* Active major bleeding requiring blood transfusion
* Other causes of thrombocytopenia such as idiopathic thrombocytopenic purpura, high clinical suspicion for heparin-induced thrombocytopenia (or other form of consumptive coagulopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Biomarkers for vascular integrity | 24 Hours
  The ratio of Angiopoietin-2 to Angiopoietin-1 is used as a measurement of vascular integrity. We will determine the change in this ratio by measuring Angiopoietin-2 (pg/mL) and Angiopoietin-1 (pg/mL) at baseline (before infusion) and 24 hours after infusion and compare between the patients receiving a unit of platelets versus the patients receiving saline.
Biomarkers for inflammation | 24 Hours
  IL-6 and TNF-alpha are commonly measured as biomarkers for inflammation. We will measure the change in concentrations (pg/mL) of IL-6 and TNF-alpha between baseline and 24 hours and compare between the population receiving a unit of platelets versus the population receiving saline.

SECONDARY OUTCOMES:
Transfusion effects on cytokines | 72 Hours
  Changes in cytokine (e.g. IL-1beta) concentrations (pg/mL) will be measured at baseline (prior to transfusion) and up to 72 hours after transfusion and compared between the population receiving a unit of platelets versus the population receiving saline.
Incidence of Serious Adverse Events | 30 days
  Each subject will be monitored for serious adverse events (e.g. death, rehospitalization) for 30 days following the platelet/saline transfusion. Outcome data will be compared between the platelet transfusion arm and the placebo arm.
Transfusion effects on coagulation | 72 Hours
  Changes in a biomarker for coagulation (prothrombin fragment 1-2) will be measured (pg/mL) at baseline (prior to transfusion) and up to 72 hours after transfusion and compared between the population receiving a unit of platelets versus the population receiving saline.
Transfusion effects on platelet number | 72 Hours
  Changes in platelet count (platelets/mm^3 blood) at baseline (prior to transfusion) and up to 72 hours after transfusion and compared between the population receiving a unit of platelets versus the population receiving saline.

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Smyth, MD PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Z, Yang F, Dunn S, Gross AK, Smyth SS. Platelets as immune mediators: their role in host defense responses and sepsis. Thromb Res. 2011 Mar;127(3):184-8. doi: 10.1016/j.thromres.2010.10.010. Epub 2010 Nov 13. PMID 21075430
- [Background] Hui P, Cook DJ, Lim W, Fraser GA, Arnold DM. The frequency and clinical significance of thrombocytopenia complicating critical illness: a systematic review. Chest. 2011 Feb;139(2):271-278. doi: 10.1378/chest.10-2243. Epub 2010 Nov 11. PMID 21071526
- [Background] Sharma B, Sharma M, Majumder M, Steier W, Sangal A, Kalawar M. Thrombocytopenia in septic shock patients--a prospective observational study of incidence, risk factors and correlation with clinical outcome. Anaesth Intensive Care. 2007 Dec;35(6):874-80. doi: 10.1177/0310057X0703500604. PMID 18084977
- [Background] Claushuis TA, van Vught LA, Scicluna BP, Wiewel MA, Klein Klouwenberg PM, Hoogendijk AJ, Ong DS, Cremer OL, Horn J, Franitza M, Toliat MR, Nurnberg P, Zwinderman AH, Bonten MJ, Schultz MJ, van der Poll T; Molecular Diagnosis and Risk Stratification of Sepsis Consortium. Thrombocytopenia is associated with a dysregulated host response in critically ill sepsis patients. Blood. 2016 Jun 16;127(24):3062-72. doi: 10.1182/blood-2015-11-680744. Epub 2016 Mar 8. PMID 26956172
- [Background] Xiang B, Zhang G, Guo L, Li XA, Morris AJ, Daugherty A, Whiteheart SW, Smyth SS, Li Z. Platelets protect from septic shock by inhibiting macrophage-dependent inflammation via the cyclooxygenase 1 signalling pathway. Nat Commun. 2013;4:2657. doi: 10.1038/ncomms3657. PMID 24150174